CLINICAL TRIAL: NCT04583943
Title: The Influence of Lifestyle Variables on Primary Dysmenorrhea; Cross-sectional Study
Brief Title: Lifestyle Influence on Primary Dysmenorrhea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, Jordan University Hospital
Other Study IDs: Questionnaire
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Menstruation Disturbances; Dysmenorrhea Primary
Keywords: Dysemnorrhea; Primary; Life style; variables
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a correlation between the effect of lifestyle and prevalence and severity of primary dysmenorrhea. We will collect data through an online questionnaire. This study is an attempt to elaborate on and clarify the prevalence and severity of primary dysmenorrhea in Jordan. This study has already been applied to other target populations therefore the purpose of this study is to establish solid numbers of dysmenorrhea prevalence in Jordan among the age group 18-25 and to exhibit a clear correlation between the lifestyle habits adopted by individuals and the intensity of dysmenorrhea present. The lifestyle factors chosen include body mass index (BMI), smoking, early menarche, prolonged menstrual flow and psychological disturbances. The significance of forming this relationship is to help raise awareness among the young generation of Jordanian women to improve on their adopted lifestyle habits in order to eventually lead to lower numbers of morbidity associated with dysmenorrhea

DETAILED DESCRIPTION:
Primary cross-sectional study. The study will be conducted in all Jordanian governorates (Amman, Irbid, Madaba, Zarqa, Balqa, Mafraq, Ajloun, Jerash, Karak, Tafileh, Maan, and Aqaba) The inclusion criteria for this study include females between the age of 18 and 25, living in Jordan only, medically free. We will not regard ethnicity and religion as part of our inclusion criteria since they are out of the scope of our research and can be specifically studied in future researches. The exclusion criteria will be; males, females beyond the age limit which is (18-25), women not living In Jordan, women having any chronic illnesses or gynecological illnesses. Moreover, participants that were unable to provide consent will be excluded from the study. The sampling technique will be simple random sampling by filling the structured self-reported online questionnaire.

A Structured self-report questionnaire which we had the approval to take it, edit it and translate it to Arabic from a research conducted in Spain(1) .It's the main tool used in this research, there will be no interviews or direct contact with the participants.

Links to the questionnaire:

Pdf version: https://drive.google.com/file/d/1K7KRLsdRbCRfdklS0wwjQv-A-Yi8le4z/view?usp=sharing Google form: https://forms.gle/8juxuMc8y3BeX9io9 Word document: https://drive.google.com/file/d/168oryAAXa1S1zvz-7KYK0p2sOob2jQxJ/view?usp=sharing The questionnaire will be sent online by using different social media panels and emails, it will be also printed out and distributed in different areas, including the university of Jordan by our team of 5th year medical students.

After data collection, data will be checked and entered. It will be analyzed using the statistical software package for the social sciences (SPSS).

We will ensure participant's privacy by not asking about their names, phone number or their address. The questionnaire will be totally anonymous. Any participant has the right to withdraw from the questionnaire at any time without repercussions.

ELIGIBILITY:
Inclusion Criteria:

Females Healthy Living in Jordan

Exclusion Criteria:

Males females beyond age group 18-25 women not living in Jordan Females with chronic medical or gynecological illness Females not able to provide consent for the study

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females between the age of 18 and 25, living in Jordan only, medically free.
Study Population: The study will be conducted in all Jordanian governorates (Amman, Irbid, Madaba, Zarqa, Balqa, Mafraq, Ajloun, Jerash, Karak, Tafileh, Maan, and Aqaba) The inclusion criteria for this study include females between the age of 18 and 25, living in Jordan only, medically free. We will not regard ethnicity and religion as part of our inclusion criteria since they are out of the scope of our research and can be specifically studied in future researches
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of primary dysmenorrhea in Jordanian females | 6 months
  Assess the prevalence of primary dysmenorrhea in Jordanian females aged 18-25
the severity of primary dysmenorrhea | 6 months
  Assess the severity of primary dysmenorrhea in Jordanian females aged 18-25
the effect of lifestyle on the prevalence and severity of primary dysmenorrhea in | 6 months
  Assess the effect of lifestyle on the prevalence and severity of primary dysmenorrhea in Jordanian females aged 18-25

SECONDARY OUTCOMES:
national recommendations to the Jordanian community regarding primary dysmenorrhea and ways to deal with this common problem. | 6 months
  Come up with national recommendations to the Jordanian community regarding primary dysmenorrhea and ways to deal with this common problem.

CONTACTS AND LOCATIONS:
Overall Officials: Al-Husban Naser, A. Professor, Principal Investigator — The University of Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Husban N, Odeh O, Dabit T, Masadeh A. The Influence of Lifestyle Variables on Primary Dysmenorrhea: A Cross-Sectional Study. Int J Womens Health. 2022 Apr 13;14:545-553. doi: 10.2147/IJWH.S338651. eCollection 2022. PMID 35444471